CLINICAL TRIAL: NCT05176028
Title: The Investigation of Acute Effects of Fascia Technique in Patients With Arthroscopic Rotator Cuff Repair: A Randomized Controlled Trial
Brief Title: Acute Effects of Fascial Release Technique in Patients With Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Çoban, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FON 2017/71
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Arthroscopic Rotator Cuff Repair
Keywords: Pain; Arthroscopic Rotator Cuff Repair; Range of Motion; Fascial Release Technique
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Hotpack, interferential current and exercise program were applied to the control group (n=15), the fascia technique was applied to the treatment group (n=15) in addition to the control group program for 2 weeks with 2 sessions per week.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): conventional physiotherapy
  Interventions: Other: conventional physiotherapy
- Intervention group (Experimental): conventional physiotherapy and fascial release
  Interventions: Other: conventional physiotherapy; Other: fascial release

INTERVENTIONS:
Other: conventional physiotherapy — For individuals of control group, hot pack applied for 20 minutes in the sitting position, Interferential Current was applied for the analgesic effect at a constant 100 Hz frequency on the anterior, posterior, superior and inferior part of the operated shoulder. By increasing the current slowly, the dosage of the current was adjusted to such a degree that the patient could tolerate it.
Other: fascial release — Fascial release technique was applied to the patients in the treatment group besides the control group program. The technique was applied to the cervical, thoracolumbar and upper extremity areas until tissue loosening and releasing were felt.
  Arms: Intervention group

SUMMARY:
This study was planned to investigate the acute effects of fascia technique on pain, range of motion, upper extremity functional level, and kinesiophobia in individuals with arthroscopic rotator cuff repair.Thirty volunteers with an arthroscopic rotator cuff repair were included to study. The individuals were randomly divided into two groups. While hot pack, interferential current and exercise program were applied to the classical physiotherapy group, the fascial release technique was applied to the treatment group in addition to the classical physiotherapy program for 2 weeks with 2 sessions per week. Individuals were assessed for pain severity by using Visual Analog Scale, range of motion by goniometer, functional level by SPADI, kinesiophobia by Tampa Kinesiophobia Scale before and after treatment and satisfaction level by using Visual Analogue Scale after treatment.

DETAILED DESCRIPTION:
Rotator cuff (RC) rupture is cause of shoulder pain, muscle weakness, decrease of shoulder range of motion (ROM), and function.The initial treatment of RC rupture is conservative treatment. The surgical option is preferred when conservative treatment is insufficient. Open, mini-open, and arthroscopic repair may be used in surgery. In the last years, mostly arthroscopic repair has preffered because of less pain, hospitalisation period, and complications than other surgical options. Postoperative rehabilitation program is important component of surgical success. The aim of this program is to decrease pain, increase ROM, and to improve function level and daily living activities of patients.Fascia is a unit connective tissue structure surrounding whole body and divided into three groups as visceral fascia, superficial fascia, and deep fascia.Fascial tissue is affected diversely due to several reasons like emotional state, injury, and surgical interventions. Inflammation because of surgery may restricts fascial tissue. Inflammation changes mechanical properties of connective tissue, cause adhesions, and finally leads to stiffness. Thereby slidings between fascial surfaces diminish, and ROM and function decrease. To release the restricted fascial tissue, several myofascial techniques are used. One of these techniques is the fascial relase technique. Myofascial techniques have effects on reducing pain, increasing ROM, and functional level. As is known, there is no study in literature for investigating the effects of fascial relase technique on pain, ROM, and function in individuals with arthroscopic RC repair. Therefore, this study was designed to investigate the acute effects of fascial release technique on pain, ROM, functional level, and kinesiophobia in patients with arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* patients undergone arthroscopic rotator cuff repair after least six weeks surgery

Exclusion Criteria:

* cervical discopathy
* shoulder osteoarthritis
* fracture or tumor of upper extremity
* adhesive capsulitis
* shoulder instability
* thoracic outlet syndrome
* neurologic or mental problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Pain severity | Before treatment, the severity of pain at rest, during activity and at night was evaluated using VAS. The starting point of the line indicated "no pain" and the end point "unbearable pain" using a 10 cm horizontal line.
  Pain is an unpleasant sensation and emotional experience.
Pain severity | After treatment, the severity of pain at rest, during activity and at night was evaluated using VAS. The starting point of the line indicated "no pain" and the end point "unbearable pain" using a 10 cm horizontal line.
  Pain is an unpleasant sensation and emotional experience.

SECONDARY OUTCOMES:
Range of motion | Before treatment, the active flexion, abduction, internal and external ROM of the individuals was evaluated using a universal goniometer in the supine position.
  Range of motion is the measurement of movement.
Range of motion | After treatment, the active flexion, abduction, internal and external ROM of the individuals was evaluated using a universal goniometer in the supine position.
  Range of motion is the measurement of movement.

OTHER OUTCOMES:
Functional level | Before treatment, SPADI was used to evaluate the functional level consists of a total of 13 items, 5 of which determine the level of pain and 8 items that determine the level of disability.
  Functional level was assessed by Shoulder Pain and Disability Index (SPADI) before and after treatment.
Fear of movement | The scale consists of 17 questions which is about the injury or re-injury in work-related activities and fear-avoidance. A 4-point Likert system is used in the scale after treatment.
  Fear of movement was evaluated by TAMPA Kinesiophobia Scale before and after treatment.
Patient satisfaction | To determine the level of satisfaction with the treatment they received, it was asked the patients to give a score between 0 (not at all satisfied) and 10 (very satisfied) using VAS after treatment.
  Patient satisfaction after treatment was assessed by VAS.
Functional level | After treatment, SPADI was used to evaluate the functional level consists of a total of 13 items, 5 of which determine the level of pain and 8 items that determine the level of disability.
  Functional level was assessed by Shoulder Pain and Disability Index (SPADI) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ertuğrul Demirdel, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Dumlupınar, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sgroi TA, Cilenti M. Rotator cuff repair: post-operative rehabilitation concepts. Curr Rev Musculoskelet Med. 2018 Mar;11(1):86-91. doi: 10.1007/s12178-018-9462-7. PMID 29399735
- [Background] Simmonds N, Miller P, Gemmell H. A theoretical framework for the role of fascia in manual therapy. J Bodyw Mov Ther. 2012 Jan;16(1):83-93. doi: 10.1016/j.jbmt.2010.08.001. Epub 2010 Sep 27. PMID 22196432
- [Background] Kain J, Martorello L, Swanson E, Sego S. Comparison of an indirect tri-planar myofascial release (MFR) technique and a hot pack for increasing range of motion. J Bodyw Mov Ther. 2011 Jan;15(1):63-7. doi: 10.1016/j.jbmt.2009.12.002. Epub 2010 Jan 27. PMID 21147420